CLINICAL TRIAL: NCT00390767
Title: A Phase I Safety, Dose Escalating Study of MultiGeneAngio in Patients With Peripheral Arterial Disease
Brief Title: Safety Study of MultiGeneAngio in Patients With Peripheral Arterial Disease (PAD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MultiGene Vascular Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGVS-MGA 001; Protocol #0504-703 (NIH RAC) (Other: NIH)
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: PAD; Claudication
Keywords: Peripheral arterial disease; Peripheral vascular disease; Claudication; Cell therapy; Gene therapy; Endothelial cells; Smooth muscle cells; Angiogenesis
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MultiGeneAngio (Experimental): Escalating doses of MultiGeneAngio
  Interventions: Biological: MultiGeneAngio

INTERVENTIONS:
Biological: MultiGeneAngio — Escalating doses of MultiGeneAngio, one dose per patient administered as one treatment, infused intra-arterially
  Other Names: MGA

SUMMARY:
The purpose of this study is to evaluate the safety and activity of increasing doses of MultiGeneAngio, a cell therapy product produced from the patient's own cells, as potential treatment for patients with peripheral arterial disease.

DETAILED DESCRIPTION:
Approximately 16 million patients worldwide (1 in 20 people over the age of 50) suffer from peripheral arterial disease(PAD). PAD is characterized by narrowing or occlusion of vessels supplying blood to the lower limbs, most often due to atherosclerosis. Symptoms of PAD include claudication that may progress to critical limb ischemia manifested by rest pain, tissue loss and gangrene, which eventually may necessitate amputation.

MultiGeneAngio is a cell therapy-based product developed for treatment of patients with PAD secondary to narrow or blocked arteries in the legs. MultiGeneAngio is composed of endothelial and smooth muscle cells that are isolated from a short vein segment stripped from the patient's arm. After isolation the cells are expanded, characterized, and gene modified by transfer of angiogenic genes.

MultiGeneAngio is a clear cell suspension injected intra-arterially at the site of blockage using a standard diagnostic catheter, in order to create and expand new collateral arteries, and thereby improve blood flow to an ischemic limb.

Comprehensive pre-clinical studies, as well as clinical experience with PAD patients suffering from claudication showed that production and administration of MultiGeneAngio was feasible and safe, as no apparent drug-related adverse events have been observed. Moreover, follow-up data of peak walking times imply a beneficial trend of this efficacy end-point. Additional follow-up data will continue to be collected to help evaluate the safety and efficacy of MultiGeneAngio.

ELIGIBILITY:
Inclusion Criteria:

* History of exercise-limiting intermittent claudication and peripheral arterial disease with symptoms in one or both legs, of at least 2 months duration with no change in symptom severity in the 2 months prior to screening.
* A Doppler-measured ankle-brachial index (ABI) of ≤0.80 or toe-brachial index (TBI) of <0.70 in at least one leg after 10 minutes of rest.
* Limitation in walking secondary to claudication with a mean peak walking time (PWT) of between 1 and 10 minutes on a standardized Gardner protocol for exercise treadmill test (ETT).
* Angiographic or equivalent anatomic evidence (MRA) of arterial occlusive disease (>70%) in the distal common femoral artery or superficial femoral artery and its branches of at least one leg within 12 months prior to screening.
* Postmenopausal (females),surgically sterile, or use adequate birth control.

Exclusion Criteria:

* Presence of significant inflow disease [defined as >50% stenosis] in the distal aorta, common or external iliac as assessed by conventional angiogram, digital subtraction angiography (DSA), or magnetic resonance angiography (MRA) performed < 1 year prior to screening.
* Critical limb ischemia, either chronic or acute ischemia manifested by rest pain, ulceration, or gangrene (Category 4 through 6 of Society for Vascular Surgery [SVS] classification [Rutherford]).
* History of malignant neoplasm (except curable non-melanoma skin malignancies).
* Renal failure (serum creatinine >2.0 mg/dL) or end-stage renal disease(requiring hemodialysis or renal replacement therapy).
* Significant hepatic disease (>3-fold elevation in ALT/AST).
* HBV or HCV carriers.
* Severe pulmonary disease (e.g. severe chronic obstructive pulmonary disease).
* Subjects with Acute Stroke within 6 months prior to screening.
* Subjects with uncontrolled diabetes mellitus.
* Specific ophthalmologic conditions that preclude retinal photography,vascular lesions of the anterior segment of the eye, proliferative retinopathy, age-related macular degeneration or intra-ocular surgery within 6 months prior to enrollment.
* Gross obesity (BMI≥40).
* Buerger's disease or other forms of inflammatory arteritis.
* Class IV congestive heart failure, as defined by the New York Heart Association or a myocardial infarction within 6 months prior to screening.
* Subject with deep vein thrombosis within 3 months prior to screening.
* Inability to complete the standardized treadmill protocol for reasons other than claudication including symptoms such as angina, dyspnea, joint pains, or excessive fatigue.
* Percutaneous intervention or surgical revascularization in the index lower limb within 6 months prior to enrollment.
* Heart angioplasty with or without stent or coronary bypass surgery within the past 6 months.
* Participation in a structured exercise treatment protocol within 30 days prior to screen testing.
* Subject is planning to participate in a structured exercise treatment protocol during the 180 days following administration of the investigational product.
* Participation in a previous gene transfer trial in which the subject received active investigational product (placebo subjects are eligible).
* Concurrent or prior participation in another clinical trial within 30 days prior to screen testing.
* Chronic use of Cox-2 inhibitors, defined as subjects needing daily use of the agent for more than 30 days prior to screening.
* Subject is taking any of the following drugs for life-threatening conditions or as part of a life-sustaining treatment: Cyclosporine (Sandimmune®),Systemic androgens/anabolic steroids, systemic corticosteroids.
* History of bleeding diathesis (e.g. hemophilia due to Factor VIII or IX deficiency).
* Pregnancy or breast-feeding.
* Uncontrolled hypertension or significant hypotension.
* Immunodeficiency states (e.g, current HIV positivity, or organ transplant recipient) or subject receiving immunosuppressive medications.
* Alcohol or other substance abuse.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The safety of MultiGeneAngio will be assessed by monitoring adverse events | Up to 15 years after treatment

SECONDARY OUTCOMES:
Improvement in PAD symptoms | Up to one year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sam L Teichman, MD, Study Director — Independent consultant
Locations (2):
- United States (2):
  - University of Michigan and VA Ann Arbor Health Systems, Ann Arbor, Michigan
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Staudacher DL, Preis M, Lewis BS, Grossman PM, Flugelman MY. Cellular and molecular therapeutic modalities for arterial obstructive syndromes. Pharmacol Ther. 2006 Jan;109(1-2):263-73. doi: 10.1016/j.pharmthera.2005.08.005. Epub 2005 Oct 21. PMID 16243400
- [Derived] Grossman PM, Mohler ER 3rd, Roessler BJ, Wilensky RL, Levine BL, Woo EY, Upchurch GR Jr, Schneiderman J, Koren B, Hutoran M, Gershstein D, Flugelman MY. Phase I study of multi-gene cell therapy in patients with peripheral artery disease. Vasc Med. 2016 Feb;21(1):21-32. doi: 10.1177/1358863X15612148. Epub 2015 Nov 19. PMID 26584888